CLINICAL TRIAL: NCT02824120
Title: Effects of Laugh Therapy Associated to Cardiopulmonary and Metabolic Rehabilitation in Ischemic Heart Disease: Randomized Clinical Trial
Brief Title: Effects of Laugh Therapy Associated to Cardiopulmonary Rehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-0124
Record Dates: First submitted 2016-02-22; First posted 2016-07-06 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Ischemic Heart Disease
Keywords: ischemic heart disease; laugh therapy
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comedy (Experimental): patients in this group will watch a comedy film that will not exceed 30 minutes
  Interventions: Other: Comedy
- Documentary (Experimental): patients in this group will watch a documentary film that will not exceed 30 minutes.
  Interventions: Other: Documentary

INTERVENTIONS:
Other: Comedy — patients will watch comedy film
  Arms: Comedy
Other: Documentary — patients will watch a documentary film
  Arms: Documentary

SUMMARY:
Laugh is more than visual and vocal behave, is always followed by a series of physiological changes, including contractions of musculoskeletal system, increase of cardiac frequency by catecholamine release and hyperventilation that promoves the increase of maximum breathing and oxygen saturation. Laugh therapy may be an alternative therapy, simple, and improve the quality of life of individuals can influence physiological and biochemical parameters of the human body.

DETAILED DESCRIPTION:
Methods: Randomized clinical trial with patients from outpatient ischemic heart disease of the Hospital de Clínicas de Porto Alegre , patients of both sexes in all regular monitoring. All patients will perform 30 minutes of stretching before film sessions. The exercises will be mild to moderate (modified Borg scale between 3 and 6).

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease diagnosis established by cardiac catheterization, with 50% lesion in at least one epicardial vessel (if the patient has had an acute coronary syndrome or have been revascularized, the event time is expected to exceed 6 months).
* Both sexes
* With availability to come to HCPA twice a week
* In conditions of entering into a cardiac rehabilitation program with exercise.

Exclusion Criteria:

* Involvement in another clinical trial.
* Presence of autoimmune disease
* Use of oral anticoagulant
* Valvulopathy with mechanical or biological cardiac prosthesis
* Presence pacemaker or implantable cardioverter
* Left bundle branch block in 12-lead ECG
* severe lung disease
* Major Depression or Bipolar Disorder
* Chronic Atrial Fibrillation
* Left ventricular dysfunction (ejection fraction <45%)
* Active infection or cancer (other than basal cell carcinoma)
* Chronic Renal Failure
* Illiteracy
* Inability to understand the consent form

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test | 48 months
  The maximum functional capacity is measured by a maximal cardiopulmonary exercise test with expired gas analysis,in the treadmill Inbramed® KT 10200 (Porto Alegre, Brazil).

SECONDARY OUTCOMES:
Quality of life Questionnaire | 48 months
  SF-36 Questionnaire of life quality

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Stein, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cortes O, Arthur HM. Determinants of referral to cardiac rehabilitation programs in patients with coronary artery disease: a systematic review. Am Heart J. 2006 Feb;151(2):249-56. doi: 10.1016/j.ahj.2005.03.034. PMID 16442885
- [Background] Briffa TG, Eckermann SD, Griffiths AD, Harris PJ, Heath MR, Freedman SB, Donaldson LT, Briffa NK, Keech AC. Cost-effectiveness of rehabilitation after an acute coronary event: a randomised controlled trial. Med J Aust. 2005 Nov 7;183(9):450-5. doi: 10.5694/j.1326-5377.2005.tb07121.x. PMID 16274344
- [Background] Yeh GY, Wood MJ, Lorell BH, Stevenson LW, Eisenberg DM, Wayne PM, Goldberger AL, Davis RB, Phillips RS. Effects of tai chi mind-body movement therapy on functional status and exercise capacity in patients with chronic heart failure: a randomized controlled trial. Am J Med. 2004 Oct 15;117(8):541-8. doi: 10.1016/j.amjmed.2004.04.016. PMID 15465501
- [Background] O'Connor GT, Buring JE, Yusuf S, Goldhaber SZ, Olmstead EM, Paffenbarger RS Jr, Hennekens CH. An overview of randomized trials of rehabilitation with exercise after myocardial infarction. Circulation. 1989 Aug;80(2):234-44. doi: 10.1161/01.cir.80.2.234. PMID 2665973
- [Background] Lu WA, Kuo CD. The effect of Tai Chi Chuan on the autonomic nervous modulation in older persons. Med Sci Sports Exerc. 2003 Dec;35(12):1972-6. doi: 10.1249/01.MSS.0000099242.10669.F7. PMID 14652490
- [Background] Martin RA. Humor, laughter, and physical health: methodological issues and research findings. Psychol Bull. 2001 Jul;127(4):504-19. doi: 10.1037/0033-2909.127.4.504. PMID 11439709
- [Background] Piegas LS, Avezum A, Pereira JC, Neto JM, Hoepfner C, Farran JA, Ramos RF, Timerman A, Esteves JP; AFIRMAR Study Investigators. Risk factors for myocardial infarction in Brazil. Am Heart J. 2003 Aug;146(2):331-8. doi: 10.1016/S0002-8703(03)00181-9. PMID 12891204
- [Background] Avezum Junior A, Feldman A, Carvalho AC, Sousa AC, Mansur Ade P, Bozza AE, Falcao Bde A, Markman Filho BM, Polanczyk CA, Gun C, Serrano Junior CV, Oliveira CC, Moreira D, Precoma DB, Magnoni D, Albuquerque DC, Romano ER, Stefanini E, Santos ES, God EM, Ribeiro EE, Brito FS, Feitosa-Filho GS, Arruda GD, Oliveira GB, Lima GG, Dohman H, Liguori IM, Costa Junior Jde R, Saraiva JF, Maia LN, Moreira LF, Santos MA, Canesin MF, Coutinho MS, Moretti AM, Ghorayeb N, Vieira NW, Dutra OP, Coelho OR, Leaes PE, Rossi PR, Andrade PB, Lemos Neto PA, Pavanello R, Costa RV, Bassan R, Esporcatte R, Miranda R, Giraldez RR, Ramos RF, Martins SK, Esteves VB, Mathias Junior W; Brazilian Society of Cardiology. [V Guideline of the Brazilian Society of Cardiology on Acute Myocardial Infarction Treatment with ST Segment Elevation]. Arq Bras Cardiol. 2015 Aug;105(2 Suppl 1):1-105. doi: 10.5935/abc.20150107. No abstract available. Portuguese. PMID 26375058
- [Background] Schmaltz HN, Southern D, Ghali WA, Jelinski SE, Parsons GA, King KM, Maxwell CJ. Living alone, patient sex and mortality after acute myocardial infarction. J Gen Intern Med. 2007 May;22(5):572-8. doi: 10.1007/s11606-007-0106-7. PMID 17443363
- [Background] Clark A, Seidler A, Miller M. Inverse association between sense of humor and coronary heart disease. Int J Cardiol. 2001 Aug;80(1):87-8. doi: 10.1016/s0167-5273(01)00470-3. PMID 11575268
- [Background] Fry WF Jr. The physiologic effects of humor, mirth, and laughter. JAMA. 1992 Apr 1;267(13):1857-8. doi: 10.1001/jama.267.13.1857. No abstract available. PMID 1545471
- [Background] Lebowitz KR, Suh S, Diaz PT, Emery CF. Effects of humor and laughter on psychological functioning, quality of life, health status, and pulmonary functioning among patients with chronic obstructive pulmonary disease: a preliminary investigation. Heart Lung. 2011 Jul-Aug;40(4):310-9. doi: 10.1016/j.hrtlng.2010.07.010. PMID 21724041
- [Background] Brutsche MH, Grossman P, Muller RE, Wiegand J, Pello, Baty F, Ruch W. Impact of laughter on air trapping in severe chronic obstructive lung disease. Int J Chron Obstruct Pulmon Dis. 2008;3(1):185-92. doi: 10.2147/copd.s2204. PMID 18488442
- [Background] Strean WB. Laughter prescription. Can Fam Physician. 2009 Oct;55(10):965-7. No abstract available. PMID 19826144
- [Background] Vlachopoulos C, Xaplanteris P, Alexopoulos N, Aznaouridis K, Vasiliadou C, Baou K, Stefanadi E, Stefanadis C. Divergent effects of laughter and mental stress on arterial stiffness and central hemodynamics. Psychosom Med. 2009 May;71(4):446-53. doi: 10.1097/PSY.0b013e318198dcd4. Epub 2009 Feb 27. PMID 19251872
- [Background] Miller M, Mangano C, Park Y, Goel R, Plotnick GD, Vogel RA. Impact of cinematic viewing on endothelial function. Heart. 2006 Feb;92(2):261-2. doi: 10.1136/hrt.2005.061424. No abstract available. PMID 16415199
- [Background] Sugawara J, Tarumi T, Tanaka H. Effect of mirthful laughter on vascular function. Am J Cardiol. 2010 Sep 15;106(6):856-9. doi: 10.1016/j.amjcard.2010.05.011. PMID 20816128
- [Background] Nasir UM, Iwanaga S, Nabi AH, Urayama O, Hayashi K, Hayashi T, Kawai K, Sultana A, Murakami K, Suzuki F. Laughter therapy modulates the parameters of renin-angiotensin system in patients with type 2 diabetes. Int J Mol Med. 2005 Dec;16(6):1077-81. PMID 16273289
- [Background] Hayashi K, Hayashi T, Iwanaga S, Kawai K, Ishii H, Shoji S, Murakami K. Laughter lowered the increase in postprandial blood glucose. Diabetes Care. 2003 May;26(5):1651-2. doi: 10.2337/diacare.26.5.1651. No abstract available. PMID 12716853
- [Background] Berk LS, Tan SA, Fry WF, Napier BJ, Lee JW, Hubbard RW, Lewis JE, Eby WC. Neuroendocrine and stress hormone changes during mirthful laughter. Am J Med Sci. 1989 Dec;298(6):390-6. doi: 10.1097/00000441-198912000-00006. PMID 2556917
- [Background] Berk LS. Studying the biology of hope: An interview with Lee S. Berk, DrPH, MPH. Interview by Sheldon Lewis. Adv Mind Body Med. 2007 Summer;22(2):28-31. PMID 20664125
- [Background] Sakuragi S, Sugiyama Y, Takeuchi K. Effects of laughing and weeping on mood and heart rate variability. J Physiol Anthropol Appl Human Sci. 2002 May;21(3):159-65. doi: 10.2114/jpa.21.159. PMID 12148458